CLINICAL TRIAL: NCT02300051
Title: Sexual Risk Behavior, Clinical and Psychopathological Aspects of Individuals With Compulsive Sexual Behavior of the Institute of Psychiatry of the General Hospital of the University of São Paulo Medical School, an Intervention Study.
Brief Title: Intervention Study for Individuals With Compulsive Sexual Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marco de Tubino Scanavino, assistant physician, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSB-2
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Compulsive Sexual Behavior
Keywords: Compulsive sexual behavior; Intervention; Short term psychodynamic group psychotherapy; Sexual addiction; Hypersexual behavior
MeSH Terms: conditions — Compulsive Sexual Behavior Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- STPGP and RPGT (Experimental): 16 weekly sessions of 90 minutes of Short-Term Psychodynamic Group Psychotherapy (STPGP) followed by 8 weekly sessions of 90 minutes of Relapse Prevention Group Therapy (RPGT)
  Interventions: Behavioral: STPGP and RPGT
- TAU (Active Comparator): Treatment as usual (TAU) will be introduced through psychiatric follow up, in which the three first visits will occur at intervals of 30 days and the followings will occur with an interval of 60 days. The medication protocol includes serotonin reuptake inhibitors (fluoxetine 20 - 80 mg/day, paroxetine 20 - 60 mg/day, sertraline 50 - 200 mg/day) or mood stabilizers (topiramate 25 - 200 mg/day, divalproex sodium (500 - 1500 mg/day, oxcarbazepine (300 - 1200 mg/day, and lamotrigine 50 - 200 mg/day).
  Interventions: Drug: TAU
- STPGP and RPGT + TAU (Experimental): Participants undergo both interventions: 1) 16 weekly sessions of 90 minutes of Short-Term Psychodynamic Group Psychotherapy (STPGP) followed by 8 weekly sessions of 90 minutes of Relapse Prevention Group Therapy (RPGT); 2)Treatment as usual (TAU) will be introduced through psychiatric follow up, in which the three first visits will occur at intervals of 30 days and the followings will occur with an interval of 60 days. The medication protocol includes serotonin reuptake inhibitors (fluoxetine 20 - 80 mg/day, paroxetine 20 - 60 mg/day, sertraline 50 - 200 mg/day) or mood stabilizers (topiramate 25 - 200 mg/day, divalproex sodium (500 - 1500 mg/day, oxcarbazepine (300 - 1200 mg/day, and lamotrigine 50 - 200 mg/day).
  Interventions: Behavioral: STPGP and RPGT; Drug: TAU

INTERVENTIONS:
Behavioral: STPGP and RPGT
  Arms: STPGP and RPGT; STPGP and RPGT + TAU
Drug: TAU
  Arms: STPGP and RPGT + TAU; TAU

SUMMARY:
The purpose of this study is compare three interventions (short-term psychodynamic psychotherapeutic group and relapse prevention group therapy vs. treatment as usual, namely, psychiatric follow up including prescription of medication vs. both interventions combined) to individuals presenting compulsive sexual behavior.

DETAILED DESCRIPTION:
We will compare three groups of patients under the three interventions, namely, (1) Short-Term Psychodynamic Group Psychotherapy (STPGP) followed by Relapse Prevention Group Therapy (RPGT) (n = 48) vs. (2) Treatment as Usual (TAU) (n = 42) vs. (3) both previous interventions combined (n = 45).

The STPGP is a 16 weekly session's group psychotherapy. Each session lasts 90 minutes. Each group will consist of around 10 participants. All the groups of STPGP will be conducted by the same psychotherapist.

The RPGT is an eight weekly therapy group. The sessions are structured and will last 90 minutes.

The medication used by those who are under TAU will be introduced through psychiatric care. Initially three visits will occur at intervals of 30 days and the followings will occur with an interval of 60 days. The medication protocol includes serotonin reuptake inhibitors (fluoxetine, paroxetine, sertraline) or mood stabilizers (topiramate, divalproex sodium, oxcarbazepine) or both type of medications combined.

All patients will be assessed on the outcomes and independent variables in the baseline (time 0); in the 25th week (time 1); and 34th week (time 2) of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. meeting the criteria for "excessive sexual drive" (ICD-10 F52.7) which corresponds to complain of an excessive sexual drive that often leads to out of control sexual behaviors AND meeting the criteria for "sex addiction" by Goodman (2001), which is characterized as a maladaptive pattern of sexual behavior leading to clinically impairment or distress as manifested in the same 12-month period by three or more of the following: tolerance (process of engaging in increasingly sexual behavior, in terms of intensity and frequency to obtain the same satisfaction than before); withdrawal (experience of abstinence, characterized by the presence of physical and/or psychological symptoms, when the behavior is diminished or discontinued); frequent sexual behavior; unsuccessful efforts to control it; many time spent in preparation for it; social or occupational activities are diminished because of it; it goes on despite negative outcomes;
2. being literate in Portuguese;
3. cognitive ability to answer self-responsive measures.

Exclusion Criteria: - individuals who met criteria for:

1. sexual preference disorders (ICD-10 F65);
2. manic or hypomanic state of bipolar disorder (ICD-10 F30.0, F31.0, 31.1, and 31.2);
3. schizophrenia, schizotypal, and delusional disorders (ICD-10 F20 - F29);
4. other mental disorders due to brain dysfunction, injury or physical disease (ICD-10 F06);
5. gender identity disorder (ICD-10 F64).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2011-02; Primary Completion 2015-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Sexual Compulsivity Scale (SCS) | Baseline, 25th and 34th week
  Changes in the total score of SCS

SECONDARY OUTCOMES:
World Health Organization Quality of Life (WHOQOL-bref) | Baseline and 25th week
  Changes in the WHOQOL-bref scores.

OTHER OUTCOMES:
Beck Depression Inventory (BDI) | Baseline and 25th week
  Changes in BDI scores
Proportion of use of condom when engaging in anal and vaginal sexual intercourse, number of casual partners | Baseline, 25th, and 34th week
  Changes in proportions of use of condom when engaging in anal and vaginal sexual intercourse, and number of casual partners reported
Beck Anxiety Inventory (BAI) | Baseline and 25th week
  Changes in BAI scores
Barratt Impulsivity Scale (BIS) 11 | Baseline, 25th, and 34th week
  Changes in BIS 11 scores
Adult Attachment Scale (AAS) | Baseline, and 25th week
  Changes in AAS scores
Knowledge and Perceptions regarding HIV transmission | Baseline, 25th week, and 34th week.
  Changes in proportion of knowledge and perceptions on HIV transmission.
Wisconsin Card Sorting Test (WCST) | Baseline, and 25th week
  Changes in scores of the neurocognitive task.
Continuous Performance Test (CPT) | Baseline, and 25th week
  Changes in scores of the neurocognitive task.
Medication adverse effect record | 25th week
  Investigation of medical records on adverse effect

CONTACTS AND LOCATIONS:
Overall Officials: Marco Scanavino, PhD, Principal Investigator — USP
Locations (1):
- Instituto de Psiquiatria do Hospital das Clínicas da Universidade de São Paulo[University of Sao Paulo General Hospital], São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Scanavino Mde T, Ventuneac A, Rendina HJ, Abdo CH, Tavares H, Amaral ML, Messina B, Reis SC, Martins JP, Gordon MC, Vieira JC, Parsons JT. Sexual Compulsivity Scale, Compulsive Sexual Behavior Inventory, and Hypersexual Disorder Screening Inventory: Translation, Adaptation, and Validation for Use in Brazil. Arch Sex Behav. 2016 Jan;45(1):207-17. doi: 10.1007/s10508-014-0356-5. Epub 2014 Oct 28. PMID 25348356
- [Background] Scanavino Mde T, Ventuneac A, Abdo CH, Tavares H, do Amaral ML, Messina B, dos Reis SC, Martins JP, Parsons JT. Compulsive sexual behavior and psychopathology among treatment-seeking men in Sao Paulo, Brazil. Psychiatry Res. 2013 Oct 30;209(3):518-24. doi: 10.1016/j.psychres.2013.01.021. Epub 2013 Feb 15. PMID 23415890
- [Background] Amaral ML, Scanavino Mde T. Severe compulsive sexual behaviors: a report on two cases under treatment. Braz J Psychiatry. 2012 Jun;34(2):213-4. doi: 10.1590/s1516-44462012000200015. No abstract available. English, Portuguese. PMID 22729419
- [Background] Scanavino Mde T, Torres RR, Abdo CH, Rego MA, Fernandez FM. Sexual compulsion and HIV transmission: a case report. Braz J Psychiatry. 2009 Jun;31(2):189-90. doi: 10.1590/s1516-44462009000200022. No abstract available. PMID 19578698
- [Background] Kafka MP. Hypersexual disorder: a proposed diagnosis for DSM-V. Arch Sex Behav. 2010 Apr;39(2):377-400. doi: 10.1007/s10508-009-9574-7. PMID 19937105
- [Background] Wainberg ML, Muench F, Morgenstern J, Hollander E, Irwin TW, Parsons JT, Allen A, O'Leary A. A double-blind study of citalopram versus placebo in the treatment of compulsive sexual behaviors in gay and bisexual men. J Clin Psychiatry. 2006 Dec;67(12):1968-73. doi: 10.4088/jcp.v67n1218. PMID 17194276
- [Background] Kaplan MS, Krueger RB. Diagnosis, assessment, and treatment of hypersexuality. J Sex Res. 2010 Mar;47(2):181-98. doi: 10.1080/00224491003592863. PMID 20358460